CLINICAL TRIAL: NCT04989933
Title: Ultrasound Guided Erector Spinae Plane Block With Two Different Volume for Open Heart Surgery: Randomized Controlled Study
Brief Title: Erector Spinae Plane Block With Two Different Volume for Open Heart Surgery
Acronym: ESP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Assoc. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AtaturkU-AnkaraCH; Asli Demir (Other: Ankara City Hospital); Ali Ahiskalioglu (Other: Ataturk University)
Record Dates: First submitted 2021-07-31; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Sternotomy Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP 20 ml (Active Comparator): Ultrasound-Guided erector spinae plane block with 20 ml of 0.25% bupivacaine
  Interventions: Procedure: Ultrasound-guided erector spinae plane block
- ESP 30 ml (Active Comparator): Ultrasound-Guided erector spinae plane block with 30 ml of 0.25% bupivacaine
  Interventions: Procedure: Ultrasound-guided erector spinae plane block

INTERVENTIONS:
Procedure: Ultrasound-guided erector spinae plane block — Ultrasound-Guided erector spinae plane block with 0.25% bupivacaine

SUMMARY:
The erector spine plane block is currently used in many surgeries to provide postoperative analgesia. It has also been used successfully in open-heart surgery for postoperative sternotomy pain. However, an ideal volume that will provide optimum analgesia has not yet been determined.

This study aims to compare the effects of ESP block administered in two different volumes on poststernotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients Undergoing Open Heart Surgery

Exclusion Criteria:

* chronic pain bleeding disorders renal or hepatic insufficiency patients on chronic non-steroidal anti-inflammatory medications emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-02 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Rescue analgesia | Post-extubation 24 hours
  Total amount of rescue analgesic